CLINICAL TRIAL: NCT05514314
Title: A Multicenter Prospective Study to Assess the Effects of Adjuvant Icotinib in EGFRm Stage I NSCLC With High-risk of Disease Recurrence After Complete Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wu Nan (Other)
Responsible Party: Sponsor-Investigator, Wu Nan, Principal Investigator, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV96
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib (Experimental): Icotinib oral 125mg tid for 2 years
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Within 4-6 weeks after surgery, Icotinib 125mg orally, TID was started for 2 years, or treatment was discontinued due to tumor recurrence or intolerance

SUMMARY:
This is a multicenter single arm study, with an aim to assess the effects of adjuvant icotinib among EGFR mutant stage I lung adenocarcinoma patients, who have high-risk pathological features of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least ≥ 18 years，and ≦ 80 years
* Lung adenocarcinoma.
* Stage I disease(IA or IB), based on TNM8 classification.
* There is at least one of the following high-risk factors:

  1. pathologically confirmed vascular invasion positive;
  2. pathologically confirmed lung adenocarcinoma containing solid or micropapillary or complex gland histology, with a percentage > 20%;
  3. pathologically confirmed invasive tumor size > 2 cm;
  4. pathologically confirmed visceral pleural involvement (T2a).
* Started adjuvant therapy in this study 4-6 weeks after complete resection without any previous antitumor therapy.
* A tumour which harbours one of the 2 EGFR mutations (Ex19del, L858R) ,without KRAS mutation
* World Health Organization performance status of 0 or 1.
* Bood routine: HB > 80g/L; ANC > 1.0x109/L; PLT > 50x109/L.Blood biochemistry： ALT and AST < 2.5 times the upper limit of normal; Crea < 1.5 times the upper limit of normal.
* Good adherence to follow-up.
* During the trial and for 3 months after the trial，Participants must be using highly effective contraceptive measures.

Exclusion Criteria:

* Prior treatment with any anticancer therapy for NSCLC (including chemotherapy, radiotherapy, immunotherapy, and EGFR-TKIs).
* Local radiotherapy.
* Patients with cancers other than NSCLC (except cured cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumors) within 5 years prior to the start of treatment in this study.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, angina pectoris beginning within the last 3 months, congestive heart failure, myocardial infarction occurring within 6 months prior to enrollment, severe arrhythmia requiring medication, liver, kidney or metabolic disease).
* Any clinical evidence suggestive of active interstitial lung disease.
* An eye inflammation or eye infection that is not fully controlled, or any condition that could lead to one of these eye conditions.
* Known human immunodeficiency virus (HIV) infection.
* Known hypersensitivity to EGFR-TKI drugs or related components.
* Mixed small cell and non-small cell cancer history.
* Substance abuse, or illnesses such as psychological or psychiatric disorders that may interfere with study compliance.
* Patients with epilepsy requiring medication (e.g. steroids or anti-epileptic drugs).
* Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to approximately 10 years
  RFS is defined as the time from the date of curative resection to the first documented recurrence or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 10 years
  OS is defined as the time from the date of randomisation until death due to any cause.
Safety and tolerability | Up to approximately 10 years
  AEs graded by CTCAE version 5.0